CLINICAL TRIAL: NCT00864331
Title: Optimization of Treatment of Advanced Nonsmall Cell Lung Cancer Using Radiotherapy and Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: International Atomic Energy Agency (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E33029
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: lung cancer; nonsmall cell lung cancer; radiation therapy; chemotherapy; Locally advanced and metastatic nonsmall cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiation; Drug Therapy; Radiotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Radiotherapy (Active Comparator): For patients in Group A (Stage IIIA or IIIB), EBRT 39 Gy in 13 daily fractions over, with no chemotherapy.
  Interventions: Radiation: radiation
- Chemotherapy and radiotherapy (Experimental): For patients in Group A (either stage IIIA or IIIB) receive a course of up to 3 cycles of chemotherapy followed by EBRT of 10 Gy in a single fraction or 16 Gy in 2 fractions 1 week apart.
  Interventions: Other: Chemotherapy and radiotherapy
- Chemotherapy (Active Comparator): For patients in Group B (either stage IIIB (wet) or IV) receive up to 3 cycles of chemotherapy, and no radiotherapy.
  Interventions: Drug: Chemotherapy
- Palliative radiotherapy and chemotherapy (Experimental): For patients in Group B (either stage IIIB (wet) or IV) receive EBRT of 10 Gy in a single fraction or 16 Gy in two fractions 1 week apart, followed by up to 3 cycles of chemotherapy.
  Interventions: Other: Palliative radiotherapy and chemotherapy

INTERVENTIONS:
Radiation: radiation — 39 Gy in 13 daily fractions of 3 Gy
  Arms: Radiotherapy
Other: Chemotherapy and radiotherapy — Chemotherapy followed by low dose palliative radiotherapy
  Arms: Chemotherapy and radiotherapy
Drug: Chemotherapy — Chemotherapy given alone
  Arms: Chemotherapy
Other: Palliative radiotherapy and chemotherapy — Low dose palliative radiotherapy followed by chemotherapy
  Arms: Palliative radiotherapy and chemotherapy

SUMMARY:
Primary objectives of the study are:

To assess the differences in survival of the two treatment options in both stage III (A and B) nonsmall cell lung cancer (NSCLC) (Study A) and Stage IIIB (wet) and stage IV NSCLC (Study B), respectively

Secondary objectives are:

To assess the differences in toxicity of two treatment options in both stage III (A and B) NSCLC (Study A) and Stage IIIB (wet) and stage IV NSCLC (Study B), and To assess the differences in Health Related Quality of Life (HRQoL) of two treatment options in both Study A and Study B

DETAILED DESCRIPTION:
To compare survival rates (median and 1-year), and toxicity of two treatment regimens in patients with locally advanced incurable NSCLC (study A), to compare survival rates (median and 1-year) of two treatment regimens in patients with locally advanced and metastatic NSCLC (study B)

To compare HRQoL and cost effectiveness of two treatment regimens in patients with locally advanced incurable NSCLC (study A), and in patients with locally advanced and metastatic NSCLC (study B) and to evaluate the effect of HRQoL assessment on QoL dimensions

ELIGIBILITY:
Study A Inclusion Criteria:

* Histologically or cytologically confirmed NSCLC
* Stage IIIA/IIIB staged with
* CT chest and upper abdomen
* Liver, renal, hematological reserve appropriate (according to "standard" institutional values)
* Brain CT and/or bone scan only if clinical symptoms request such investigation
* Performance status KPS 60-90
* No second cancer except skin non-melanoma
* No previous treatment
* Patient must be contactable for follow-up
* Patient to be able to start treatment within 2 weeks from randomization (institutional confirmation needed)
* Life expectancy > 3 months
* Patient must be able and willing to give informed consent, and fill in questionnaires

Study A Exclusion Criteria:

* Stage III B "wet" (existing pleural effusion , but not necessarily cytologically verified)
* RT field > 200 cm2
* Pregnancy

Study B Inclusion Criteria:

* KPS 60-90
* Stage IV and Stage III B (existing pleural effusions , but not necessarily cytologically verified)
* Histologically or cytologically confirmed
* CT staged disease (thorax and possible upper abdomen)
* No second cancer except skin non-melanoma
* Liver, renal, haematological reserve appropriate (according to "standard" institutional values)
* No previous treatment
* Patient must be contactable for follow-up
* Patient must be able and willing to give informed consent and fill in questionnaires
* Patient to be able to start treatment within 2 weeks from randomization (institutional confirmation needed)
* Life expectancy > 3 months

Study B Exclusion Criteria:

* Brain metastasis (brain CT and/or MRI not needed, unless symptoms exist - clinically indicated)
* RT field > 200 cm2
* Pregnancy
* A-P separation too large to be adequately treated with 60-Co (?)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2008-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Survival | 1 year

SECONDARY OUTCOMES:
To assess the differences in toxicity of two treatment options in both stage III (A and B) NSCLC (Study A) and Stage IIIB (wet) and stage IV NSCLC (Study B) | 1 year
To assess the differences in Health Related Quality of Life (HRQoL) of two treatment options in both Study A and Study B | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Elena Fidarova, MD, Principal Investigator — International Atomic Energy Agency
Locations (13):
- Instituto de Radiomedicine, Santiago, Chile
- Affiliated Hospital of Ning Xia Medical College, Department of Radiation Oncology, Yinchuan, China
- University of Zagreb Faculty of Medicine, Zagreb, Croatia
- Misr Oncology Center (MOC), Cairo, Egypt
- Tata Memorial Centre (TMC) Department of Atomic Energy (DAE), Mumbai, India
- General Hospital Kuala Lumpur, Institute of Radiotherapy and Oncology, Kuala Lumpur, Malaysia
- Sir Paul Boffa Hospital, Floriana, Malta
- Ministère de la Santé, Institut National d'Oncologie Sidi Mohamed Ben Abdellah, Rabat, Morocco
- Nuclear Medicine Oncology and Radiotherapy Institute, Islamabad, Pakistan
- Instituto Oncológico National, Panama City, Panama
- Instituto Nacional de Enfermadades Neoplasicas Depto. De Radioterapia, Lima, Peru
- University of Witwatersrand Johannesburg Hospital Dept of Radiation Oncology, Johannesburg, South Africa
- Institut de la Sante Publique, Institut National de Cancer Salah Azaiz, Tunis, Tunisia

REFERENCES:
- [Derived] Jeremic B, Fidarova E, Sharma V, Faheem M, Ameira AA, Nasr Ben Ammar C, Frobe A, Lau F, Brincat S, Jones G. The International Atomic Energy Agency (IAEA) randomized trial of palliative treatment of incurable locally advanced non small cell lung cancer (NSCLC) using radiotherapy (RT) and chemotherapy (CHT) in limited resource setting. Radiother Oncol. 2015 Jul;116(1):21-6. doi: 10.1016/j.radonc.2015.06.017. Epub 2015 Jul 7. PMID 26163093